CLINICAL TRIAL: NCT07241533
Title: A Clinical Efficacy Study of Asiaticoside for Treating Overweight/Obesity
Brief Title: Asiaticoside for Treating Overweight/Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-710
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Overweight , Obesity
Keywords: obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — asiaticoside

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Participants take Asiaticoside tablets 60mg tid for 12 weeks
  Interventions: Drug: Asiaticoside tablets

INTERVENTIONS:
Drug: Asiaticoside tablets — Asiaticoside tablets 60mg tid for 12 weeks

SUMMARY:
Centella asiatica is a traditional herbal medicine widely used in China and Southeast Asia for treating various conditions. Preclinical studies have shown that madecassic acid glycosides, including asiaticoside and madecassoside, can significantly reduce body weight gain, adipose tissue mass, and serum triglyceride levels in high-fat diet-induced obese mice. These compounds also improve hepatic steatosis and insulin resistance. This exploratory, interventional study aims to evaluate the clinical efficacy of orally administered asiaticoside tablets in adults with overweight or obesity.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older, male or female.
* Overweight or obesity, defined as a body mass index (BMI) of 24.0-45.0 kg/m².
* Able and willing to provide written informed consent.

Exclusion Criteria:

* Active pulmonary tuberculosis, malignant tumors, human immunodeficiency virus (HIV) infection, or other severe infectious or immunocompromising conditions.
* Severe liver injury (AST or ALT > 3 times the upper limit of normal) or severe renal dysfunction/end-stage renal disease (eGFR < 30 mL/min/1.73 m²).
* Severe cardiovascular diseases, including angina pectoris, myocardial infarction, or stroke within the past 6 months.
* Severe gastrointestinal disorders, or a history of gastrointestinal surgery within the past year.
* Secondary causes of obesity, including Cushing's syndrome, primary hypothyroidism, hypothalamic obesity, acromegaly; or drug-induced obesity (e.g., antipsychotics, glucocorticoids).
* Currently receiving other anti-obesity treatments, a previous history of bariatric surgery, or a >5% reduction in body weight within the past 3 months.
* Current smoker or habitual smoker within the past 3 months.
* type 1 or type 2 diabetes mellitus or currently taking hypoglycemic medications.
* Pregnancy or planning pregnancy, or breastfeeding.
* Unable to complete a 3-month follow-up due to health conditions or relocation.
* Participation in any clinical study within the past 4 weeks.
* Other conditions considered by investigators as unsuitable for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in Metabolic Rate | Baseline to Week 4
  Metabolic rate will be assessed using indirect calorimetry in a metabolic chamber (whole-room indirect calorimetry) at baseline and Week 4 after taking Asiaticoside tablets.
Change in Body Weight | Baseline to Week 12
  Body weight will be measured using a calibrated digital scale at baseline and Week 12 after taking Asiaticoside tablets.

SECONDARY OUTCOMES:
Change in Body Mass Index (BMI) | Baseline to Week 12
  Body mass index (BMI) will be calculated as weight (kg) divided by height squared (m²). This outcome assesses changes in BMI from baseline to Week 12.
Change in Body Fat Percentage | Baseline to Week 12
  Body fat percentage will be evaluated using dual-energy X-ray absorptiometry (DEXA) at baseline and Week 12 after taking Asiaticoside tablets.
Change in waist circumference | From baseline to Week 12
  Waist circumference will be measured using standardized anthropometric methods at baseline and Week 12 after taking Asiaticoside tablets.
Change in Blood Pressure | Baseline to Week 12
  Systolic and diastolic blood pressure will be assessed at baseline and Week 12 after taking Asiaticoside tablets.
Change in Lipid profile | Baseline to Week 12
  Fasting lipid profile (TC, TG, LDL-C, HDL-C) will be assessed at baseline and Week 12 after taking Asiaticoside tablets.
Change in HbA1c | Baseline to Week 12
  Hemoglobin A1c will be assessed at baseline and Week 12 after taking Asiaticoside tablets.
Change in Insulin Sensitivity (HOMA-IR) | Baseline to Week 12
  HOMA-IR will be calculated at baseline and Week 12 after taking Asiaticoside tablets. HOMA-IR is calculated using the following equation: HOMA-IR = fasting plasma glucose in mmol/L×fasting insulin in μU/ml/22.5.
Change in Leptin Levels | Baseline to Week 12
  Serum leptin levels will be measured at baseline and Week 12 after taking Asiaticoside tablets.
Change in High-Sensitivity C-Reactive Protein (hs-CRP) | Baseline to Week 12
  High-sensitivity C-reactive protein levels will be measured at baseline and Week 12 after taking Asiaticoside tablets.
Change in Liver Fat Content | Baseline to Week 12
  Liver fat content will be represented by the Controlled Attenuation Parameter (CAP) with FibroScan at baseline and Week 12 after taking Asiaticoside tablets.
Change in Liver Stiffness | Baseline to Week 12
  Liver stiffness will be represented by Liver Stiffness Measurement (LSM) with FibroScan at baseline and Week 12 after taking Asiaticoside tablets.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: After publication.
Access Criteria: IPD and supporting information will be avaible to researchers upon reasonable request (e.g. with a practical and meaningful research proposal).